CLINICAL TRIAL: NCT02113345
Title: The Relationship Between Metamemory and Memory in Old Age
Acronym: M&Mresearch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 082010Deb
Record Dates: First submitted 2014-03-12; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Mild Cognitive Impairment
Keywords: metamemory; memory; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counseling (Experimental): Metamemory Cognitive Intervention
  Interventions: Behavioral: Metamemory Cognitive Intervention

INTERVENTIONS:
Behavioral: Metamemory Cognitive Intervention — Metamemory Cognitive Intervention

SUMMARY:
The purpose of this research is to explore the relationship of metamemory and memory of elders and to evaluate the effectiveness of a metamemory cognitive intervention on elders with mild cognitive impairment and low memory self-efficacy.

DETAILED DESCRIPTION:
There are 3 studies in the present research. Study 1 is a reliability and validity study of the Chinese Metamemory Scales. Study 2 is a cross-sectional study to explore the relationship between metamemory and memory of elders encountered in Hong Kong primary health care setting.Study 3 is an Effectiveness Study of Metamemory Cognitive Intervention on elders with mild cognitive impairment and low memory self-efficacy.

This research has the following aims and hypotheses:

Research Aims:

1. To evaluate the reliability and validity of the Chinese Metamemory Scales
2. To explore the relationship between metamemory and memory of elders
3. To evaluate the effectiveness of a metamemory cognitive intervention on Mild Cognitive Impairment (MCI) elders who have low memory self-efficacy

Research Hypotheses:

Study 1: The Chinese Metamemory Scales will show acceptable psychometric properties.

Study 2: There is a positive correlation between metamemory (subjective memory) and memory (objective memory) and this relationship is mediated by stereotyped beliefs about memory ageing.

Study 3: Comparing to Control Group, the Intervention Group will yield the following expected results:

1. There is an improvement in objective memory measures post-training.
2. There is an improvement in subjective memory measures post-training.
3. There is an improvement in mood measures post-training.

ELIGIBILITY:
Inclusion Criteria:

* Study 1:

Participants are Chinese elderly of age 65 or above and they speak Cantonese as their primary language. They are to be recruited from a convenience sample of clients who are without cognitive problems and are attending service in the Elderly Health Centres (EHC) of the Elderly Health Service of the Department of Health, Hong Kong Special Administrative Region Government (HKSARG).

* Study 2:

In addition to the inclusion criteria of Study 1, EHC members with confirmed dementia, suspected dementia, and suspected MCI will also be invited to participate in Study 2. However, confirmed demented clients and suspected demented clients must show their capacity to appraise by passing Quality of Life Appraisal Inventory (CapQOL) (Wong, J.G.W.S. et al., 2005) before they are accepted to the Study. All clients are recruited upon consent.

* Study 3:

Suspected MCI participants of Study 2 with below average memory self-efficacy assessed to have MCI (according to operational definition) will be invited and recruited to Study 3 upon consent. In the present research, MCI is defined operationally according to prior local studies and determined with reference to the educational level-adjusted cutoff scores of Chinese Mini Mental Status Examination (CMMSE) and Abbreviated version of Memory Inventory for the Chinese combined (Lam, L. C.W. & et al., 2005; Lam, L.C.W. & et al., 2008).

Exclusion Criteria:

* The presence of currently active medical conditions potentially affecting cognition e.g. vitamin B12 deficiency, hypothyroidism, chronic alcoholism, delirium, and active psychiatric disorders e.g. schizophrenia
* Other conditions that might affect cognitive competency e.g. aphasia, severe visual or hearing impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Objective Memory Measures | Baseline, post-intervention at week 16
  change from baseline in Hong Kong List Learning Test, 2nd Edition (HKLLT, Chan, A.S., 2006) for verbal episodic memory
Objective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in Figure Recognition of Memory Assessment Scale (MAS, Williams, 1991) for visual episodic memory
Objective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in Category Verbal Fluency Test (CVFT, categories to be chosen with reference to local studies by published by Chiu, H.F.K. et al., 1997 and Mok et al., 2004) for semantic memory
Objective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in Digit Span and Visual Spatial Span from (MAS, Williams, 1991) for verbal and visual memory working memory
Objective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in Event-based and Time-based Tasks for prospective memory (tasks to be developed with reference to the recommendations of Wilson, B.A. & et al., 2008)

SECONDARY OUTCOMES:
Subjective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in the Chinese version of Memory Self-efficacy Scale (MSE, Frequency of Forgetting-10 Scale, Zelinski and Gilewski, 2004)
Subjective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in Chinese versions of the Abbreviated version of Memory Inventory for the Chinese (AMIC, Lam, Linda, C. W. & et al., 2005)
Subjective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in Chinese versions of the Anxiety about Memory (AM, a subscale of the Memory Functioning Questionnaire, Gilewski, Zelinski & Schaie, 1990, for Study 1 only)
Subjective Memory Measures | Baseline, post-intervention at week 16
  Change from baseline in Chinese versions of the Stereotypes about Memory Aging (SMA, Fort & Gana, 2009)

CONTACTS AND LOCATIONS:
Overall Officials: Debbie SK Chow, Principal Investigator — The University of Hong Kong
Locations (1):
- Research Site, Hong Kong, Hong Kong